CLINICAL TRIAL: NCT03518723
Title: Effect and Feasibility of Non-linear Periodized Resistance Training in People With Chronic Obstructive Pulmonary Disease: a Randomized Controlled Multicenter Trial
Brief Title: Effect and Feasibility of Non-linear Periodized Resistance Training in People With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other); Radboud University Medical Center (Other); Merem Pulmonary Rehabilitation Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NLPRT-RCT
Record Dates: First submitted 2018-04-13; First posted 2018-05-08 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Disease; Chronic Obstructive
Keywords: Muscle dysfunction
MeSH Terms: conditions — Lung Diseases | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Prospective, assessor-blind, parallel-group randomized controlled multicenter trial with a pre- and post-intervention design
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors will be masked to group allocation. The participants will be given repeated instructions not to reveal their group allocation to the outcome assessors. In case of failure in keeping the outcome assessor masked (i.e, a patient reveals his/her group allocation), a second trained outcome assessor will be available.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-linear Periodized Resistance Training (Experimental): The objective of the Non-linear Periodized Resistance Training (NLPRT) program is to increase muscle strength as well as muscle endurance. The NLPRT program will over the 8 week intervention period target several different aspects of limb muscle function, by alternating the intensity and volume of the exercises.
  Progression of exercise is symptom dependent and will be based on Borg CR-10 ratings (dyspnea, muscle fatigue and exertion).
  All exercises will be performed using exercise equipment that are available at each included center.
  All sessions are supervised and conducted by local professionals using a group format, with approximately 2-4 participants per group.
  Interventions: Other: Non-linear Periodized Resistance Training
- Resistance Training (Active Comparator): The primary objective of the Resistance training (RT) group is to increase muscular strength. The RT program will be performed in line with current guidelines that are recommended for increasing muscular strength in patients with COPD.
  Progression of exercise is performance dependent and will be based on the previous 2 sessions.
  All exercises will be performed using exercise equipment that are available at each included center.
  All sessions are supervised and conducted by local professionals using a group format, with approximately 2-4 participants per group.
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: Non-linear Periodized Resistance Training — 8 week non-linear periodized resistance training intervention, 3 sessions per week, 60 minutes per session
  Arms: Non-linear Periodized Resistance Training
Other: Resistance training — 8 week resistance training intervention, 3 sessions per week, 60 minutes per session
  Arms: Resistance Training

SUMMARY:
This study aims at improving the knowledge about resistance training for people with COPD. Resistance training is an important part of pulmonary rehabilitation when the goal is to improve muscular endurance and strength. The study will evaluate the effects and the feasibility of two resistance training programs for people with COPD using a parallel group design. One program will include a larger day-to-day variation (i.e. non-linear periodization) and the progression will be guided by ratings of dyspnea, muscle fatigue, and exertion. The other program will follow the established guidelines for resistance training for people with COPD. The programs will be evaluated for effects regarding muscular endurance, strength, intramuscular adaptions, functional preformance, dyspnea, and health related quality of life. The programs will also be evaluated for feasibility regarding the duration of training sessions, attendance rates, adverse events, and participant satisfaction. The hypothesis is that the non-linear periodization group will have superior effects and that feasibility aspects will be similar between groups.

ELIGIBILITY:
Inclusion Criteria:

* FEV1/FVC ratio < 70% postbronchodilator
* FEV1 <80% of the predicted normal value postbronchodilator

Exclusion Criteria:

* Clinical evidence of asthma, cardiovascular diseases, and/or neuromuscular diseases that are unstable and/or that may contribute to exercise limitation
* Other contraindications to exercise
* Currently participating in a structured exercise or pulmonary rehabilitation program or been involved in pulmonary rehabilitation in the past 6 months
* Experienced a COPD exacerbation and/or change in medication dosage/frequency in the past 6 weeks

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline dynamic maximal endurance at week 9 | Baseline and week 9
  Maximal limb muscle endurance measured using resistance training machines or free weights. Reported as the number of repetitions at 45% of the baseline one repetition maximum.
Change from baseline dynamic maximal strength at week 9 | Baseline and week 9
  Maximal limb muscle strength measured using resistance training machines or free weights. Reported as one repetition max in kg.

SECONDARY OUTCOMES:
Change from baseline static maximal endurance at week 9 | Baseline and week 9
  Maximal limb muscle endurance measured using a computerized dynamometer or strain gauge. Reported in seconds maintaining 60% of the isometric maximal voluntary contraction.
Change from baseline static maximal strength at week 9 | Baseline and week 9
  Maximal limb muscle strength measured using a computerized dynamometer or strain gauge. Reported in Nm
Change from baseline unsupported upper limb test (UULEX) at week 9 | Baseline and week 9
  The UULEX is a progressive test where the participants will be asked to a raise plastic bar from the hip to the UULEX eight-level chart with a cadence of 30 movements per minute. If a patient reaches the highest level, the plastic bar will be replaced by a heavier one every minute. There are five different bar weights (0.2, 0.5, 1, 1.5, 2 Kg) and participants will continue on the highest level until symptom limitation. Results are reported in seconds.
Change from baseline endurance shuttle walk test (ESWT) at week 9 | Baseline and week 9
  The ESWT is a derivative of the Incremental shuttle walk test (ISWT), where patients walk for as long as possible at a predetermined percentage of maximum walking performance as assessed by the ISWT on a 10 meter course. Reported in seconds to termination of the test or total meters walked.
Change from baseline 60 seconds sit to stand test (60STS) at week 9 | Baseline and week 9
  During the 60STS, participants will be instructed to fully stand up and sit down as fast as possible, as many times as possible within 60 seconds. Arms will be held fold across the chest with feet remaining in full contact with the floor. Reported as the number of repetitions performed within 60 seconds.
Change From Baseline Chronic Respiratory Questionnaire Self-Administered Standardized Format (CRQ-SAS) Total Scores at week 9 | Baseline and week 9
  The CRQ-SAS is a self-administered questionnaire which consist of 20 items across four domains: dyspnea (5 items), fatigue (4 items), emotional function (7 items), and mastery (4 items). Participants rates their experience on a 7-point scale in response to each item ranging from 1 (maximum impairment) to 7 (no impairment). Individual items are equally weighted, and total score ranges from 20 to 140 (20 maximum impairment, 140 no impairment).
Change From Baseline Chronic Respiratory Questionnaire Self-Administered Standardized Format (CRQ-SAS) dyspnea Domain Scores at week 9 | Baseline and week 9
  Domain scores are calculated as the mean of all items (5) within the dyspnea domain. Participants rates their experience on a 7-point scale in response to each item ranging from 1 (maximum impairment) to 7 (no impairment). Individual items are equally weighted, and total score ranges from 7 to 35 (7 maximum dyspnea, 35 no dyspnea).
Number of responders | Week 9
  The total amount of responders i.e. defined as a response over the known minimal detectable change/or minimal important difference for included test(s) will be determined and compared.
Attendance rate | Week 1 up to 8
  Attendance rate will be evaluated by calculating the number of attended sessions divided by total number of sessions for each participant
Duration of exercise sessions | Week 1 up to 8
  Mean time in minutes of exercise sessions
Satisfaction rate | Week 9
  Participant satisfaction with the exercise regimens will be recorded by adapting an existing patient satisfaction questionnaire. Participants rate their satisfaction on 7 items each with a 5 point likert scale. Results using the total score (0-35, higher score indicating higher satisfaction).
Proportion of drop-outs | Week 9
  Proportion of participants that don't complete the intervention
Adverse Events rate | Week 1 up to 8
  Occurrence of any adverse events. An adverse event rate will be calculated for each patient as the total number of sessions during which any adverse events occurred divided by the total number of attended sessions.
Adverse Events stratified by severity | Week 1 up to 8
  The severity of the adverse events will be assessed and rated into four different categories: 1) minor and temporary, 2) serious symptoms (potential risk of severe injury or life threatening), 3) manifest injury or disease, and 4) death. Presented in factual numbers for each group.
Change from baseline muscle fiber size at week 9 | Baseline and week 9
  The tissue sample obtained from the vastus lateralis muscle will be examined with morphometric analyses to determine cross-sectional fiber area. Reported in square micrometers.
Change from baseline proportion of slow and fast subtypes of contractile myosin heavy chain isoforms in fibers at week 9 | Baseline and week 9
  The tissue sample obtained from the vastus lateralis muscle will be examined with immunohistochemistry techniques to categorize fiber types.
Change from baseline oxidative (citrate synthase (CS), EC 4.1.3.7) enzyme activities at week 9 | Baseline and week 9
  The tissue sample obtained from the vastus lateralis muscle will be examined to demonstrate enzyme activities. Reported in micromol/min/g tissue.
  [Time Frame: Baseline and week 9] The tissue sample obtained from the vastus lateralis muscle will be examined by histochemistry to demonstrate enzyme activities. Reported in micromol/min/g tissue.
Change from baseline glycolytic (lactate dehydrogenase (LDH), EC 1.1.1.27) enzyme activities at week 9 | Baseline and week 9
  The tissue sample obtained from the vastus lateralis muscle will be examined to demonstrate enzyme activities. Reported in micromol/min/g tissue.
Change from baseline capillarization (capillary density) at week 9 | Baseline and week 9
  The tissue sample obtained from the vastus lateralis muscle will be examined with morphometric analysis to determine capillary density, estimated as the total number of capillaries per millimeter squared muscle cross-section.
Change from baseline capillarization (capillaries to fiber) at week 9 | Baseline and week 9
  The tissue sample obtained from the vastus lateralis muscle will be examined with morphometric analysis to determine the number of capillaries around fibers including all capillaries in contact with each muscle fiber.
Change from baseline capillarization (capillaries relative to fiber area) at week 9 | Baseline and week 9
  The tissue sample obtained from the vastus lateralis muscle will be examined with morphometric analysis to determine the number of capillaries around each fiber relative to its cross-sectional area.

CONTACTS AND LOCATIONS:
Overall Officials: Andre Nyberg, PhD, Principal Investigator — Umeå University
Locations (3):
- Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Canada
- Merem Pulmonary Rehabilitation Centre, Hilversum, Netherlands
- Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frykholm E, Klijn P, Saey D, van Hees HWH, Stal P, Sandstrom T, Sorlin A, Maltais F, Nyberg A. Effect and feasibility of non-linear periodized resistance training in people with COPD: study protocol for a randomized controlled trial. Trials. 2019 Jan 3;20(1):6. doi: 10.1186/s13063-018-3129-y. PMID 30606240